CLINICAL TRIAL: NCT06571864
Title: AL Amyloidosis and Anti-CD38-Daratunumab
Acronym: AL38
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DARA_01
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD38 (Experimental): Daratumumab is intravenously given at the dose of 16 mg/kg weekly for 8 weeks, then every two weeks for 8 more times, and lastly monthly until the 52nd week (8 more administrations)
  Interventions: Drug: Anti-CD38 Monoclonal Antibody

INTERVENTIONS:
Drug: Anti-CD38 Monoclonal Antibody — Anti-CD38 Monoclonal Antibody: Daratumumab is intravenously given at the dose of 16 mg/kg weekly for 8 weeks, then every two weeks for 8 more times, and lastly monthly until the 52nd week (8 more administrations)

SUMMARY:
AL Amyloidosis and anti-CD38

DETAILED DESCRIPTION:
AL amyloidosis is a systemic disorder characterized by progressive multiorgan failure and premature death. While autologous stem cell transplantation (ASCT) is considered the standard therapy, eligibility is limited, and excludes a substantial proportion of patients. Recent guidelines recommend daratumumab-based regimens for these patients, but, particularly for cases with severe renal involvement, optimal treatment remains a challenge.

This study explore the efficacy of daratumumab monotherapy in patients with histologically proven severe renal involvement who are ineligible for ASCT

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by AL amyloidosis
* Patients who were ineligible for high dose therapy and bone marrow transplantation due to age and/or frailty score.

Exclusion criteria:

- Diagnosis of AL amyloidosis not biospy proven

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
organ responses were defined according to the updated International Society of Amyloidosis criteria | "through study completion, an average of 1 year".

CONTACTS AND LOCATIONS:
Overall Officials: Dario Roccatello, Principal Investigator — ASL Città di Torino, Torino, IT
Locations (1):
- San Giovanni Bosco Hospital, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No